CLINICAL TRIAL: NCT03120052
Title: Defining Components of Physical Therapy Achieving Maximum Function After Total Knee Replacement
Brief Title: Physical Therapy Components for Maximum TKR Outcome
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Patricia Franklin, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: NIH 1 R01 AR071048-01; 1R01AR071048-01 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis; Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this study is to identify what Physical Therapy care components are associated with the best patient-reported functional outcome after Total Knee Replacement (TKR) surgery. The investigators are specifically looking at outcomes at 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled to undergo an elective, unilateral primary total knee replacement due to knee osteoarthritis
* Will receive outpatient PT from a participating physical therapist.
* Agree to record their exercise and activity for specific time points in the study.

Exclusion Criteria:

* Total knee replacement scheduled for indications other than OA (e.g., fracture, malignancy, infection, or revision or prior implant)
* The inability to obtain informed consent due to cognitive conditions.
* Non-English speakers as the materials used in this project have not yet been tested with non-English speakers
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients electing total knee replacement at one of participating PT sites.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Differences in overall functional gain at 6 months | 6 month follow-up
  Differences in pre-operative to 6 month post -operative functional gain, using the SF-36 Physical Component Summary (PCS) Score by physical therapy regimen.

SECONDARY OUTCOMES:
Differences in knee specific functional gain at 6 months | 6 month follow-up
  Differences in pre-operative to 6 month post-operative functional gain, using the Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living (ADL) by physical therapy regimen.
Differences in knee performance measures at 6 months | 6 month follow-up
  Differences in pre-operative to 6-month post -operative knee performance measures using the Physical Therapy Performance Measures (includes a 5 minute stair climbing exercise, a 6 minute walking exercise and a sit to stand exercise) by physical therapy regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D Franklin, MD, MBA, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical SChool, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franklin PD, Li W, Ayers DC. The Chitranjan Ranawat Award: functional outcome after total knee replacement varies with patient attributes. Clin Orthop Relat Res. 2008 Nov;466(11):2597-604. doi: 10.1007/s11999-008-0428-8. PMID 18810570
- [Background] Han AS, Nairn L, Harmer AR, Crosbie J, March L, Parker D, Crawford R, Fransen M. Early rehabilitation after total knee replacement surgery: a multicenter, noninferiority, randomized clinical trial comparing a home exercise program with usual outpatient care. Arthritis Care Res (Hoboken). 2015 Feb;67(2):196-202. doi: 10.1002/acr.22457. PMID 25220488
- [Background] Freburger JK, Holmes GM, Ku LJ, Cutchin MP, Heatwole-Shank K, Edwards LJ. Disparities in post-acute rehabilitation care for joint replacement. Arthritis Care Res (Hoboken). 2011 Jul;63(7):1020-30. doi: 10.1002/acr.20477. PMID 21485020
- [Background] Naylor J, Harmer A, Fransen M, Crosbie J, Innes L. Status of physiotherapy rehabilitation after total knee replacement in Australia. Physiother Res Int. 2006 Mar;11(1):35-47. doi: 10.1002/pri.40. PMID 16594314
- [Background] Westby MD, Brittain A, Backman CL. Expert consensus on best practices for post-acute rehabilitation after total hip and knee arthroplasty: a Canada and United States Delphi study. Arthritis Care Res (Hoboken). 2014 Mar;66(3):411-23. doi: 10.1002/acr.22164. PMID 24023047
- [Background] Peter WF, Jansen MJ, Hurkmans EJ, Bloo H, Dekker J, Dilling RG, Hilberdink W, Kersten-Smit C, de Rooij M, Veenhof C, Vermeulen HM, de Vos RJ, Schoones JW, Vliet Vlieland TP; Guideline Steering Committee - Hip and Knee Osteoarthritis. Physiotherapy in hip and knee osteoarthritis: development of a practice guideline concerning initial assessment, treatment and evaluation. Acta Reumatol Port. 2011 Jul-Sep;36(3):268-81. PMID 22113602
- [Background] Ebert JR, Munsie C, Joss B. Guidelines for the early restoration of active knee flexion after total knee arthroplasty: implications for rehabilitation and early intervention. Arch Phys Med Rehabil. 2014 Jun;95(6):1135-40. doi: 10.1016/j.apmr.2014.02.015. Epub 2014 Mar 3. PMID 24602550
- [Background] Ruiz D Jr, Koenig L, Dall TM, Gallo P, Narzikul A, Parvizi J, Tongue J. The direct and indirect costs to society of treatment for end-stage knee osteoarthritis. J Bone Joint Surg Am. 2013 Aug 21;95(16):1473-80. doi: 10.2106/JBJS.L.01488. PMID 23965697
- [Background] Ong KL, Lotke PA, Lau E, Manley MT, Kurtz SM. Prevalence and Costs of Rehabilitation and Physical Therapy After Primary TJA. J Arthroplasty. 2015 Jul;30(7):1121-6. doi: 10.1016/j.arth.2015.02.030. Epub 2015 Feb 28. PMID 25765130
- [Background] Lingard EA, Berven S, Katz JN; Kinemax Outcomes Group. Management and care of patients undergoing total knee arthroplasty: variations across different health care settings. Arthritis Care Res. 2000 Jun;13(3):129-36. PMID 14635286
- [Background] Roos EM. Effectiveness and practice variation of rehabilitation after joint replacement. Curr Opin Rheumatol. 2003 Mar;15(2):160-2. doi: 10.1097/00002281-200303000-00014. PMID 12598806
- [Background] Oatis CA, Li W, DiRusso JM, Hoover MJ, Johnston KK, Butz MK, Phillips AL, Nanovic KM, Cummings EC, Rosal MC, Ayers DC, Franklin PD. Variations in Delivery and Exercise Content of Physical Therapy Rehabilitation Following Total Knee Replacement Surgery: A Cross-Sectional Observation Study. Int J Phys Med Rehabil. 2014;Suppl 5:002. doi: 10.4172/2329-9096.S5-002. Epub 2014 Apr 22. PMID 26594649
- [Background] Peter WF, Nelissen RG, Vlieland TP. Guideline recommendations for post-acute postoperative physiotherapy in total hip and knee arthroplasty: are they used in daily clinical practice? Musculoskeletal Care. 2014 Sep;12(3):125-31. doi: 10.1002/msc.1067. Epub 2014 Feb 4. PMID 24497426
- [Background] Dejong G, Horn SD, Smout RJ, Tian W, Putman K, Gassaway J. Joint replacement rehabilitation outcomes on discharge from skilled nursing facilities and inpatient rehabilitation facilities. Arch Phys Med Rehabil. 2009 Aug;90(8):1284-96. doi: 10.1016/j.apmr.2009.02.009. PMID 19651262
- [Background] DeJong G, Tian W, Smout RJ, Horn SD, Putman K, Smith P, Gassaway J, Davanzo JE. Use of rehabilitation and other health care services by patients with joint replacement after discharge from skilled nursing and inpatient rehabilitation facilities. Arch Phys Med Rehabil. 2009 Aug;90(8):1297-305. doi: 10.1016/j.apmr.2008.12.029. PMID 19651263
- [Background] Fritz JM, Hunter SJ, Tracy DM, Brennan GP. Utilization and clinical outcomes of outpatient physical therapy for medicare beneficiaries with musculoskeletal conditions. Phys Ther. 2011 Mar;91(3):330-45. doi: 10.2522/ptj.20090290. Epub 2011 Jan 13. PMID 21233306
- [Background] Artz N, Dixon S, Wylde V, Beswick A, Blom A, Gooberman-Hill R. Physiotherapy provision following discharge after total hip and total knee replacement: a survey of current practice at high-volume NHS hospitals in England and wales. Musculoskeletal Care. 2013 Mar;11(1):31-8. doi: 10.1002/msc.1027. Epub 2012 Jul 9. PMID 22778023
- [Background] Pozzi F, Snyder-Mackler L, Zeni J. Physical exercise after knee arthroplasty: a systematic review of controlled trials. Eur J Phys Rehabil Med. 2013 Dec;49(6):877-92. Epub 2013 Oct 30. PMID 24172642
- [Background] Rosal MC, Ayers D, Li W, Oatis C, Borg A, Zheng H, Franklin P. A randomized clinical trial of a peri-operative behavioral intervention to improve physical activity adherence and functional outcomes following total knee replacement. BMC Musculoskelet Disord. 2011 Oct 7;12:226. doi: 10.1186/1471-2474-12-226. PMID 21981909
- [Background] Petterson SC, Mizner RL, Stevens JE, Raisis L, Bodenstab A, Newcomb W, Snyder-Mackler L. Improved function from progressive strengthening interventions after total knee arthroplasty: a randomized clinical trial with an imbedded prospective cohort. Arthritis Rheum. 2009 Feb 15;61(2):174-83. doi: 10.1002/art.24167. PMID 19177542
- [Background] Bade MJ, Stevens-Lapsley JE. Early high-intensity rehabilitation following total knee arthroplasty improves outcomes. J Orthop Sports Phys Ther. 2011 Dec;41(12):932-41. doi: 10.2519/jospt.2011.3734. Epub 2011 Sep 30. PMID 21979411
- [Background] Minns Lowe CJ, Barker KL, Dewey M, Sackley CM. Effectiveness of physiotherapy exercise after knee arthroplasty for osteoarthritis: systematic review and meta-analysis of randomised controlled trials. BMJ. 2007 Oct 20;335(7624):812. doi: 10.1136/bmj.39311.460093.BE. Epub 2007 Sep 20. PMID 17884861
- [Background] Skoffer B, Dalgas U, Mechlenburg I. Progressive resistance training before and after total hip and knee arthroplasty: a systematic review. Clin Rehabil. 2015 Jan;29(1):14-29. doi: 10.1177/0269215514537093. Epub 2014 Jul 3. PMID 24994766
- [Background] Zech A, Hendrich S, Pfeifer K. Association Between Exercise Therapy Dose and Functional Improvements in the Early Postoperative Phase After Hip and Knee Arthroplasty: An Observational Study. PM R. 2015 Oct;7(10):1064-1072. doi: 10.1016/j.pmrj.2015.04.008. Epub 2015 Apr 16. PMID 25892356
- [Background] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888
- [Background] Spangehl MJ. Is It Time for Telerehabilitation to Go Mainstream? J Bone Joint Surg Am. 2015 Jul 15;97(14):e55. doi: 10.2106/JBJS.O.00540. No abstract available. PMID 26178897
- [Background] Kramer JF, Speechley M, Bourne R, Rorabeck C, Vaz M. Comparison of clinic- and home-based rehabilitation programs after total knee arthroplasty. Clin Orthop Relat Res. 2003 May;(410):225-34. doi: 10.1097/01.blo.0000063600.67412.11. PMID 12771834
- [Background] NIH Consensus Panel. NIH Consensus Statement on total knee replacement December 8-10, 2003. J Bone Joint Surg Am. 2004 Jun;86(6):1328-35. doi: 10.2106/00004623-200406000-00031. No abstract available. PMID 15173310
- [Background] Goldstein MS, Scalzitti DA, Craik RL, Dunn SL, Irion JM, Irrgang J, Kolobe TH, McDonough CM, Shields RK. The revised research agenda for physical therapy. Phys Ther. 2011 Feb;91(2):165-74. doi: 10.2522/ptj.20100248. Epub 2010 Dec 17. No abstract available. PMID 21169424
- [Background] White NT, Delitto A, Manal TJ, Miller S. The American Physical Therapy Association's top five choosing wisely recommendations. Phys Ther. 2015 Jan;95(1):9-24. doi: 10.2522/ptj.20140287. Epub 2014 Sep 15. No abstract available. PMID 25223237
- [Background] Franklin PD, Allison JJ, Ayers DC. Beyond joint implant registries: a patient-centered research consortium for comparative effectiveness in total joint replacement. JAMA. 2012 Sep 26;308(12):1217-8. doi: 10.1001/jama.2012.12568. No abstract available. PMID 23011710